CLINICAL TRIAL: NCT03117595
Title: Combined Spinal Epidural Analgesia in Labour: A Comparison of Two Intrathecal Regimens of Single Shot Spinal
Brief Title: CSE for Labour Analgesia: A Comparison of Two Intrathecal Regimens
Acronym: SSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarah Beckley (Other)
Responsible Party: Sponsor-Investigator, Sarah Beckley, Senior Registrar and Diplomate, Dept of Anaesthesia, General Hospital, Gbagada Lagos, Nigeria, Lagos State Health Service Commission
Organization: Lagos State Health Service Commission (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAS/17/03
Record Dates: First submitted 2017-04-09; First posted 2017-04-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain
Keywords: Single Shot Spinal; Intrathecal narcotics; Morphine; Fentanyl; Labour Analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: 2 groups that would remain with the randomly picked intervention throughout the study duration
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: a double blinded study. The participant and the Physician giving the treatment who would also evaluate the participant during the duration of the study are masked. However, the Assistant who is in charge of the randomization process and has the code and so would prepare the drugs is not blinded. The non-blinded Assistant would be available to break the code in the event of any adverse reactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BF (Active Comparator): Interventions: Intrathecal administration -Bupivacaine 2.5mg (0.5ml) + Fentanyl 25mcg (0.5ml) + 1ml sterile water in one shot Ephedrine 3-5mg in aliquots in the event of hypotension Promethazine 12.5 - 25mg in the event of vomiting or significant pruritus naloxone 2mcg/kg in the event of respiratory distress
  Interventions: Drug: Bupivacaine-fentanyl
- BFM (Active Comparator): Interventions: Intrathecal administration - Bupivacaine 2.5mg (0.5ml) + fentanyl 25mcg (0.5ml) + 0.25mg morphine (0.25ml) + 0.75ml sterile water in one shot ephedrine 3-5mg in aliquots for hypotension Promethazine 12.5 - 25mg for vomiting or significant pruritus Naloxone 2mcg/kg in the event of respiratory distress
  Interventions: Drug: Bupivacaine-fentanyl morphine

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — Dosages as previously written
  Arms: BF
Drug: Bupivacaine-fentanyl morphine — Dosage as previously written
  Arms: BFM

SUMMARY:
Analgesia in labour is not readily available in many parts of Sub-Saharan Africa. The overall cost of Epidural services in terms of human personnel and financial implication makes this inaccessible to many women in labour. Thus, a cheaper, less technically demanding and easier option that can produce as much satisfaction for the parturient and would allow her participate in the second stage of labour by being able to bare down is being studied.

The Single Shot Spinal (SSS) would provide pain relief in these women however its draw back is its time limitation as the option of a top up is not available.

Two regimen of drug options would be considered using opioids. These would be compared to see how well they are able to provide analgesia in women who hitherto have had vaginal birth. Their onset, duration of action and possible side effects would be compared.

NULL HYPOTHESIS: Single Shot Spinal with Bupivacaine Fentanyl (BF) cannot provide a statistically significant difference in labour analgesia in comparison with Bupivacaine Fentanyl Morphine (BFM) ALTERNATE HYPOTHESIS: Single Shot Spinal with BF can provide a statistically significant difference in labour in comparison with BFM

DETAILED DESCRIPTION:
A double blinded randomized study comparing 2 intrathecal mixtures for labour analgesia.

94 multiparous parturients in active labour who have given informed consent would be recruited into the study. They would be randomly allocated into 2 groups using simple random sampling. An Assistant would know the code and prepare the intrathecal solutions.

Baseline vitals would be taken and patient's pain score noted. Due protocol would be followed and a combined spinal epidural sited but with the epidural not activated until the effect of the spinal wears off.

Routine monitoring would be done and various parameters and indices noted. Where the effect of the spinal lasts the duration of labour thus no need to activate the epidural, this would also be noted.

Data would be analysed using Statistical Package of Social Sciences (SPSS) version 20.

ELIGIBILITY:
Inclusion Criteria:

* Parturients in active labour >4cm dilatation
* American Society of Anesthesiologists (ASA) classification I and II

Exclusion Criteria:

* Significant co-morbidities like uncontrolled hypertension or diabetes
* Maternal hemorrhage with hypotension
* Significant bleeding/clotting disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Time to First painless contraction (TFC) | time zero to first painless contraction estimated 15 minutes
  This is the onset of action of the drugs. The time duration from the initiation of the block at time zero to the point where there is significant drop in the Numerical Rating Scale (NRS) to 2 or less
Time to First Request for Analgesia (TFA) | Time zero till NRS > 6 estimated 180 minutes
  This is the duration of action of the block. Time from initiation of the block to time the pain score is up to 6 or more. It is expected that after onset of the block (TFC) the pain would first become negligible or absent and after a period of time, it would gradually increase as the drug wears off. If the pain becomes moderate at a NRS of 6 or the patient requests for analgesia, the time would be noted and the epidural would be activated.

SECONDARY OUTCOMES:
Delivery before TFA or delivery after TFA | duration of labour estimated 180 minutes
  Qualitative variable. determines if rescue analgesia was needed (if the epidural needed to be activated) or if the spinal was adequate for the duration of labour
Maternal Satisfaction | up to 300 minutes
  Parturients perception of if analgesia was Adequate, Inadequate or Not Sure
Side effects | up to 180 minutes
  Presence of side effects like respiratory depression, pruritus, or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Olaniyi Oladapo, MBBS,FMCA, FWACS, Study Chair — School of Anaesthetic Studies, Health Service Commission, Lagos State
Locations (1):
- Lagos Island Maternity Centre, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Minty RG, Kelly L, Minty A, Hammett DC. Single-dose intrathecal analgesia to control labour pain: is it a useful alternative to epidural analgesia? Can Fam Physician. 2007 Mar;53(3):437-42. PMID 17872679
- [Background] Lee BB, Ngan Kee WD, Hung VY, Wong EL. Combined spinal-epidural analgesia in labour: comparison of two doses of intrathecal bupivacaine with fentanyl. Br J Anaesth. 1999 Dec;83(6):868-71. doi: 10.1093/bja/83.6.868. PMID 10700784
- [Background] Hess PE, Vasudevan A, Snowman C, Pratt SD. Small dose bupivacaine-fentanyl spinal analgesia combined with morphine for labor. Anesth Analg. 2003 Jul;97(1):247-52, table of contents. doi: 10.1213/01.ane.0000066520.30763.b8. PMID 12818975